CLINICAL TRIAL: NCT07004985
Title: The Effect of Reinforcement With Kahoot and Google Forms on Midwifery Students' Success and Motivation in the Normal Birth and Postpartum Period Course and Their Opinions
Brief Title: Gamified and Form-Based Reinforcement in Midwifery Education: A Quasi-Experimental Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Antalya Bilim University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2024\993; Antalya Bilim University (Other: Antalya Bilim University, Faculty of Health Sciences, Department of Midwifery)
Record Dates: First submitted 2025-05-27; First posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Educational Reinforcement; Midwifery Education; Student Motivation; Academic Achievement; Gamification in Health Education
Keywords: Kahoot; Google Forms; Educational intervention; Academic performance; Normal Birth and Postpartum Period course

STUDY DESIGN:
Masking Description: Participants and investigators are aware of the group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kahoot Group (Experimental): This group will receive digital reinforcement through gamified quizzes using the Kahoot platform. Following the theoretical portion of the "Normal Birth and Postpartum Period" course, participants will engage in four interactive quiz sessions on Kahoot, each consisting of 25 multiple-choice questions. The reinforcement aims to enhance engagement, motivation, and knowledge retention through real-time feedback and competition elements.
  Interventions: Behavioral: Kahoot Reinforcement; Behavioral: Google Forms Reinforcement
- Google Forms Group (Experimental): This group will receive digital reinforcement through structured multiple-choice quizzes delivered via Google Forms. After the theoretical lessons of the "Normal Birth and Postpartum Period" course, students will complete four quiz sessions using Google Forms, each including 25 questions. This reinforcement method is designed to support repetition, comprehension, and motivation through reflective practice and immediate feedback.
  Interventions: Behavioral: Kahoot Reinforcement; Behavioral: Google Forms Reinforcement

INTERVENTIONS:
Behavioral: Kahoot Reinforcement — Students in this group will complete four interactive reinforcement sessions using the Kahoot platform, following the theoretical content of the "Normal Birth and Postpartum Period" course. Each session includes 25 multiple-choice questions delivered in a gamified format, with real-time feedback and scoring. The intervention aims to increase motivation, focus, and retention of knowledge.
Behavioral: Google Forms Reinforcement — Students in this group will complete four structured reinforcement sessions using Google Forms, after participating in the same theoretical course content. Each session consists of 25 multiple-choice questions, delivered in a self-paced online format. The intervention supports repetition and reflection, aiming to improve academic performance and motivation.

SUMMARY:
This quasi-experimental study aims to evaluate the effect of reinforcement using Kahoot (a gamification tool) and Google Forms (an interactive quiz platform) on the academic achievement and motivation of midwifery students enrolled in the "Normal Birth and Postpartum Period" course. The study involves two intervention groups: one using Kahoot and the other using Google Forms. A total of 39 third-year midwifery students will participate. Academic success will be measured through pre- and post-tests, motivation levels through a validated motivation scale, and qualitative feedback will be obtained through student opinion forms. The study seeks to explore how different digital reinforcement tools affect learning outcomes and student engagement in midwifery education.

DETAILED DESCRIPTION:
This quasi-experimental study investigates the impact of two different digital reinforcement tools-Kahoot and Google Forms-on third-year midwifery students' academic performance and motivation in the "Normal Birth and Postpartum Period" course. A total of 39 students will be assigned to two groups based on the last digit of their student ID number: even-numbered students will form the Kahoot group (n=19), and odd-numbered students will form the Google Forms group (n=20).

Both groups will receive the same theoretical course content over a 7-week period, followed by different reinforcement strategies. The Kahoot group will complete gamified multiple-choice quizzes via the Kahoot platform, while the Google Forms group will answer the same questions using structured forms. The reinforcement process includes 4 quiz sessions in one day, each with 25 questions, and will be followed by a pre-test, post-test, and administration of the Motivated Strategies for Learning Questionnaire.

Academic achievement will be assessed through a standardized 25-item multiple-choice test developed and validated by academic experts. Motivation levels will be measured using the Turkish version of the Instructional Materials Motivation Survey (IMMS), based on the ARCS model (Attention, Relevance, Confidence, Satisfaction). In addition, student opinions will be collected through Likert-type and open-ended questions regarding their experiences with the reinforcement tools.

The goal is to determine whether different forms of digital reinforcement influence student performance and engagement, and to identify students' perspectives on their learning experience. All participants will voluntarily participate and the study will be conducted in accordance with ethical standards.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the "Normal Birth and Postpartum Period" course during the 2024-2025 academic year
* Being a third-year midwifery student at Antalya Bilim University
* Having access to a smartphone
* Voluntarily agreeing to participate in the study

Exclusion Criteria:

* Absence on the day of data collection
* Declining to participate in the study
* Not completing both pre- and post-tests
* Technical inability to access Kahoot or Google Forms platforms

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-01-20 (Actual); Study Completion 2025-06-25 (Estimated)

PRIMARY OUTCOMES:
Change in Academic Achievement Score | Pre-test at Week 1, Post-test at Week 6
  Assessed through a 25-question multiple-choice test specifically developed for the "Normal Birth and Postpartum Period" course. Scores range from 0 to 100.
Change in Motivation Level | Before intervention (Week 1) and after intervention (Week 6)
  Measured using the Turkish-adapted version of the Instructional Materials Motivation Survey (IMMS). Scores range from 33 to 165.

SECONDARY OUTCOMES:
Student Opinions on Digital Reinforcement Tools | Week 7
  Collected via a Likert-scale and open-ended questionnaire designed to assess student experiences with Kahoot and Google Forms.

CONTACTS AND LOCATIONS:
Overall Officials: Seda Serhatlıoğlu, Doctorate, Principal Investigator — Antalya Bilim University, Faculty of Health Sciences, Department of Midwifery
Locations (1):
- Antalya, Döşemealtı, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code